CLINICAL TRIAL: NCT01283997
Title: A Phase II Study of Minocycline vs. Placebo to Prevent Treatment Induced Neuropathy in Multiple Myeloma
Brief Title: Prevention of Treatment Induced Neuropathy in Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-0022; NCI-2011-00247 (Registry Identifier: NCI CTRP); 1P01CA124787-01 (NIH)
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Myeloma
Keywords: Multiple Myeloma; Neuropathy; Peripheral Nerve Function; Touch Detection Threshold; Nerve Damage; Thalidomide; Bortezomib; Velcade; Minocycline; Dynacin; Minocin; Minocin PAC; Myrac; Solodyn
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): 1 dose on first day of induction therapy, then every 12 hours for 10 weeks.
  Interventions: Other: Placebo
- Minocycline Group (Experimental): 200 mg orally for 1 dose, then 100 mg orally every 12 hours for 10 weeks.
  Interventions: Drug: Minocycline

INTERVENTIONS:
Other: Placebo — One pill by mouth on Day 1. Staring on Day 2, 2 times a day (every 12 hours) by mouth for 10 weeks.
  Arms: Placebo Group
Drug: Minocycline — 200 mg by mouth for 1 dose, then 100 mg by mouth every 12 hours for 10 weeks.
  Other Names: Dynacin; Minocin; Minocin PAC; Myrac; Solodyn
  Arms: Minocycline Group

SUMMARY:
The goal of this clinical research study is to see if Minocin® (minocycline) can help to control nerve damage that causes numbness and tingling in the hands and feet (neuropathy) in patients receiving thalidomide and/or bortezomib.

DETAILED DESCRIPTION:
Neuropathy is one of the side effects that occurs in some patients who receive thalidomide and/or bortezomib. Usually it is mild and sometimes improves or goes away when the thalidomide or bortezomib treatment is stopped. However, in some patients, the numbness and tingling remains even after the treatment is stopped. It can make it difficult for patients to feel objects with their hands, or to feel the ground under their feet. This can lead to difficulty with tasks such as buttoning clothes or writing, as well as difficulty walking.

Minocycline is designed to help prevent inflammation of the nerves, which can stop the nerve cells from dying.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. Participants in the 2 groups will receive standard education from the study staff about the signs and symptoms of neuropathy. If you are assigned to Group A, you will take a placebo (pills that look like the study drug but do not contain any active ingredients) once on Day 1. Staring on Day 2, you will take the pills 2 times a day (every 12 hours), for 10 weeks. If you are assigned to Group B you will take a larger dose of minocycline 1 time by mouth on the day you start therapy on this study, and then a smaller dose of minocycline by mouth every 12 hours for 10 weeks. Minocycline can be taken with or without food, but it needs to be taken with liquid. No matter which group you are assigned to, you will receive thalidomide and/or bortezomib according to the standard schedule. Neither you nor your doctor nor any of the clinic or research staff will know which medication (placebo or minocycline) you are receiving. Only the pharmacist who gives you the medication will know. If there is any serious concern for your safety because of the medication you might be receiving, your doctor will be told which medication you are receiving.

Study Visits:

One (1) time a week during Weeks 1-9, you will complete the symptom questionnaire. This questionnaire may be done in person or by phone.

Before you begin each new cycle of multiple myeloma therapy for 10 weeks, the following tests and procedures will be performed:

* You will have a physical exam.
* Your complete medical history will be recorded, and you will be asked about any drugs you may be taking.
* Your performance status will be recorded.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.
* Blood (about 4 teaspoons) will be drawn to test for certain cytokines.
* You will have a nerve function test.
* You will complete the questionnaire that has questions about unusual sensations you may experience in your arms, legs, hands, and feet and problems these sensations may cause for you.
* You will complete the symptom questionnaire that has questions about pain, fatigue, nausea, disturbed sleep, difficulty remembering, mood, work, and enjoyment of life.
* You will complete a questionnaire that asks about high likely you are to doze off or fall asleep while doing certain activities. This should take about 2-3 minutes.
* You will be asked about any side effects you may have experienced.

End-of-Study Visit:

Once you have completed the study medication (minocycline or placebo) after Week 10, you will be asked to return for an end-of-study visit:

* You will have a physical exam.
* Your complete medical history will be recorded, and you will be asked about any drugs you may be taking.
* Your performance status will be recorded.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.
* Blood (about 4 teaspoons) will be drawn to test for certain cytokines.
* You will have a nerve function test and a neuro-cognitive test.
* You will complete the questionnaire that has questions about unusual sensations you may experience in your arms, legs, hands, and feet and problems these sensations may cause for you.
* You will complete the symptom questionnaire that has questions about pain, fatigue, nausea, disturbed sleep, difficulty remembering, mood, work, and enjoyment of life.
* You will complete a questionnaire that asks about high likely you are to doze off or fall asleep while doing certain activities. This should take about 2-3 minutes.
* You will be asked about any side effects you may have experienced.

If intolerable side effects occur, or if thalidomide and/or bortezomib for the myeloma is stopped, you will be taken off study.

This is an investigational study. Minocycline is commercially available and FDA approved for use in other diseases, such as infections caused by bacteria. Minocycline is not FDA approved for the treatment of neuropathy. In neuropathy, it is currently being used in research only. Up to 142 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed English speaking patients with symptomatic multiple myeloma who have received 1 or fewer treatment cycles of thalidomide or bortezomib, and who will receive thalidomide and/or twice-weekly schedule bortezomib as part of induction therapy for their multiple myeloma
2. Age greater than or equal to 18 years
3. Able to render informed consent and to follow protocol requirements
4. Women must be postmenopausal (no menstrual period for a minimum of 1 year) or if they are of childbearing potential they must agree to use adequate birth control measures (e.g. abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, implantable or injectable contraceptives or surgical sterilization during the study
5. Men must agree to use adequate birth control measures (e.g. abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, implantable or injectable contraceptives or surgical sterilization) during the study.

Exclusion Criteria:

1. Hypersensitivity to tetracyclines
2. Poorly controlled or advanced diabetes mellitus (hemoglobin A1c >/= 8 %)
3. Women who are pregnant or nursing
4. Patients with peripheral neuropathy of >/= grade 2 by CTCAE v4.0.
5. Have a history of alcohol or substance abuse within the preceding 6 months that, in the opinion of the investigator, may increase the risks associated with study participation or study agent administration, or may interfere with interpretation of results
6. Currently have any known malignancy other than multiple myeloma, or have a history of malignancy within the previous 5 years, with the exception of basal cell or squamous cell carcinoma of the skin that has been fully excised with no evidence of recurrence
7. Have current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease
8. Inability to use interactive voice recognition software due to physical limitations (e.g. hearing impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2011-01-25 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheeba K. Thomas, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 79 Participants signed consent
Groups:
- Placebo Group: Participants received a placebo of one dose on the first day of induction therapy for multiple myeloma, then doses every 12 hours for 10 weeks.
- Minocycline Group: Participants received minocycline 200 mg orally for 1 dose, then 100 mg orally every 12 hours for 10 weeks beginning at initiation of induction therapy for multiple myeloma
Period: Overall Study
Arm/Group | Placebo Group | Minocycline Group
Started | 39 | 40
Completed | 23 | 23
Not Completed | 16 | 17
Not completed — Physician Decision | 8 | 10
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Physically unable to continue | 0 | 1
Not completed — Progressive disease | 1 | 0
Not completed — Other | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Placebo Group: Participants received one pill by mouth on Day 1. Staring on Day 2, 2 times a day (every 12 hours) by mouth for 10 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Minocycline Group | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 27 | 51
  >=65 years | 15 | 13 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 23 | 24 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 35 | 36 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 28 | 30 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 39 | 40 | 79

OUTCOME MEASURES:

1. Primary Outcome: The Difference Between Touch Detection Thresholds From the Sensorimotor Evaluation at Baseline and After 10 Weeks of Induction Therapy.
Description: Touch detection thresholds are determined using the up/down method with calibrated von Frey monofilaments,
  Starting with a 0.5mN force, the von Frey monofilament is applied for approximately 1 sec. If the subject fails to detect the stimulus, then the next higher force von Frey monofilament is applied. When the subject detects the presence of the stimulus, the next lower von Frey is administered. The up/down test sequence continues until the same force filament is detected for three additional applications. The force of that filament is then assigned as the touch threshold
Time Frame: baseline and week 10
Measure: Mean (Standard Deviation); unit: mN
Arm/Group | Placebo Group | Minocycline Group
Number analyzed (Participants) | 17 | 19
mN
  Fingertips | 0.00 (0.25) | 0.06 (0.28)
  Thenar Eminence | 0.08 (0.26) | 0.13 (0.27)
  Volar Forearm | 0.09 (0.36) | -0.03 (0.44)
Statistical Analysis 1: Comparison: Placebo Group vs Minocycline Group; Difference in the measurements for touch by the fingertip; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.13 to 0.24]
Statistical Analysis 2: Comparison: Placebo Group vs Minocycline Group; Difference in the measurements for touch by the palm; Test type: Other; p = 0.60, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.13 to 0.23]
Statistical Analysis 3: Comparison: Placebo Group vs Minocycline Group; Difference in the measurements for touch by the forearm; Test type: Other; p = 0.37, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.40 to 0.15]

2. Secondary Outcome: Change in the Mean Value of Patient-reported MD Anderson Symptom Inventory for Multiple Myeloma (MDASI-MM) Numbness Scores From Baseline to Week 10 Post Treatment.
Description: Participants reported the severity of two cognitive symptoms numbness on a 0-10 scale, with 0 being 'not present' and 10 being 'as bad as you can imagine': Higher mean scores indicate more severe symptoms.
Time Frame: baseline and week 10
Population: Participants with quantitative sensory testing (QST) done a week prior to the start of their minocycline treatment and with corresponding QST at week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Group | Minocycline Group
Number analyzed (Participants) | 21 | 20
score on a scale | 1.38 (2.36) | 0.65 (1.79)
Statistical Analysis 1: Comparison: Placebo Group vs Minocycline Group; Difference in Numbness severity at baseline and week 10; Test type: Other; p = 0.56, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.73, 95% CI 2-sided [-2.06 to 0.59]

ADVERSE EVENTS:
Time Frame: From the first dose through 330 days after the last dose of study medication
Arm/Group | Placebo Group | Minocycline Group
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 15/39 | 12/40
Other Adverse Events (participants affected / at risk) | 39/39 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Group (N=39) | Minocycline Group (N=40)
Elevated SGPT (Investigations) | 1 | 0
Elevated serum myeloma protein (Investigations) | 6 | 10
Elevated urinary protein (Renal and urinary disorders) | 2 | 1
Elevated serum and urine protein (Renal and urinary disorders) | 1 | 1
Pain - back (Musculoskeletal and connective tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Abnormal serum and urine (Renal and urinary disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Elevated LDH (Investigations) | 1 | 0
Elevated serum total protein (Investigations) | 1 | 0
Elevated serum myeloma protein (Renal and urinary disorders) | 1 | 0
Fungal pharyngitis (Infections and infestations) | 1 | 0
Phosphatase, elevated serum proteins (Investigations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Elevated serum and urinary myeloma protein (Renal and urinary disorders) | 5 | 7
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Group (N=39) | Minocycline Group (N=40)
Anemia (Blood and lymphatic system disorders) | 21 | 24
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 | 0 — Abnormal CBC, cell-shape and size
Hematuria (Renal and urinary disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 1 — Back spasm
Edema Limbs (General disorders) | 3 | 5 — Calf swelling
Constipation (Gastrointestinal disorders) | 9 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blood and lymphatic system disorders - Other, specify (Investigations) | 2 | 0 — Decreased Monocyte
Investigations - Other, specify (Investigations) | 1 | 0 — Decreased S-Chloride
Blood and lymphatic system disorders - Other, specify (Investigations) | 2 | 1 — Decreased eosinophil
Anemia (Blood and lymphatic system disorders) | 2 | 1
Lymphocyte count decreased (Investigations) | 2 | 0
Depression (Psychiatric disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 1
Dry eye (Eye disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Generalized edema (General disorders) | 4 | 2
Creatinine increased (Investigations) | 3 | 2
Alkaline phosphatase increased (Investigations) | 10 | 8
Aspartate aminotransferase increased (Investigations) | 13 | 9
Alanine aminotransferase increased (Investigations) | 5 | 3
Investigations - Other, specify (Investigations) | 1 | 2 — Elevated absolute neutrophil count
Investigations - Other, specify (Injury, poisoning and procedural complications) | 6 | 8 — elevated BUN
Blood bilirubin increased (Investigations) | 3 | 2
Investigations - Other, specify (Investigations) | 5 | 3 — elevated carbon dioxide
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 10 | 14
Investigations - Other, specify (Investigations) | 0 | 1 — Elevated LD2
Investigations - Other, specify (Investigations) | 0 | 1 — Elevated LFT
Investigations - Other, specify (Investigations) | 1 | 1 — Elevated S Chloride
Investigations - Other, specify (Investigations) | 0 | 1 — Elevated S Guanine
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Investigations - Other, specify (Investigations) | 11 | 11 — Elevated S. myeloma proteins
Investigations - Other, specify (Investigations) | 1 | 0 — Elevated S. total protein
Thyroid stimulating hormone increased (Investigations) | 0 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 9 | 7 — Elevated U. myeloma protein
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Investigations - Other, specify (Investigations) | 0 | 1 — Elevated granulocyte
Investigations - Other, specify (Investigations) | 1 | 3 — Elevated immature granulocyte
Fatigue (General disorders) | 5 | 6
Fever (General disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
: - Hypercalcemia (Metabolism and nutrition disorders) | 3 | 2
Cholesterol high (Investigations) | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 2 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 4 | 4
Hypertension (Vascular disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 | 12
Hyponatremia (Metabolism and nutrition disorders) | 5 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 8 | 9
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 4
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 1 — Hypoproteinemia
Hypotension (Vascular disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 0 — Jitters
Lip pain (Gastrointestinal disorders) | 0 | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 | 2 — decrease eosinophil
Lymphocyte count decreased (Investigations) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 8
Amnesia (Nervous system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 17 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 | 1 — Pneumonia
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 4
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 2
Oral pain (Gastrointestinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Superficial thrombophlebitis (Vascular disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 | 2 — Elevated mean platelet volume
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 | 0 — Elevated mean platelet count
Investigations - Other, specify (Investigations) | 1 | 0 — Elevated metamyelocyte
Investigations - Other, specify (Investigations) | 0 | 1 — Elevated metamyelocyte percent
Investigations - Other, specify (Investigations) | 1 | 3 — Elevated monocyte percent
Investigations - Other, specify (Investigations) | 1 | 0 — Elevated neutrophil
Investigations - Other, specify (Investigations) | 2 | 2 — Elevated neutrophil percent
Investigations - Other, specify (Investigations) | 0 | 1 — Elevated neutrophil percent and ANC
Proteinuria (Renal and urinary disorders) | 2 | 2
Eye Pain (Eye disorders) | 0 | 1
Pain (General disorders) | 7 | 8
Investigations - Other, specify (Investigations) | 1 | 0 — reduced chloride
Neutrophil count decreased (Investigations) | 1 | 0
Investigations - Other, specify (Investigations) | 0 | 1 — reduced serum CO2
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0 — Ca oxalate crystals
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 1 — Urinary casts

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT01283997/Prot_SAP_000.pdf